# THE OHIO STATE UNIVERSITY AUTHORIZATION TO USE PERSONAL HEALTH INFORMATION IN RESEARCH

**Title of the Study:** OSU 19305 (NCI #10317): A Pilot Study of Nivolumab in Combination with Decitabine and Venetoclax in TP53-mutated Acute Myeloid Leukemia **Protocol Number:** IRB# 2019Y0039

Principal Investigator: Dr. Alice Mims

| Subject Name |
|--------------|
|--------------|

Before researchers use or share any health information about you as part of this study, The Ohio State University is required to obtain your authorization. This helps explain to you how this information will be used or shared with others involved in the study.

- The Ohio State University and its hospitals, clinics, health-care providers, and researchers are required to protect the privacy of your health information.
- You should have received a Notice of Privacy Practices when you received health care services here. If not, let us know and a copy will be given to you. Please carefully review this information. Ask if you have any questions or do not understand any parts of this notice.
- If you agree to take part in this study your health information will be used and shared with others involved in this study. Also, any new health information about you that comes from tests or other parts of this study will be shared with those involved in this study.
- Health information about you that will be used or shared with others involved in this study may include your research record and any health care records at The Ohio State University. For example, this may include your medical records, x-rays, or laboratory results. Psychotherapy notes in your health records (if any) will not, however, be shared or used. Use of these notes requires a separate, signed authorization.

Please read the information carefully before signing this form. Please ask if you have any questions about this authorization, the university's Notice of Privacy Practices or the study before signing this form.

#### Those Who May Use, Share, and Receive Your Information as Part of This Study

• Researchers and staff at The Ohio State University will use, share, and receive your personal health information for this research study. Authorized Ohio State staff not involved in the study may be aware that you are participating in a research study and have access to your information. If this study is related to your medical care, your study-related information may be placed in your permanent hospital, clinic, or physician's office records.

- Those who oversee the study will have access to your information, including the following:
  - Members and staff of The Ohio State University's Institutional Review Boards, including the Western Institutional Review Board
  - The Ohio State University Office of Responsible Research Practices
  - University data safety monitoring committees
  - The Ohio State University Office of Research.
- Your health information may also be shared with federal and state agencies that have oversight of the study or to whom access is required under the law. These may include the following:
  - Food and Drug Administration
  - Office for Human Research Protections
  - National Institutes of Health
  - Ohio Department of Job and Family Services.
- These researchers, companies and/or organization(s) outside of The Ohio State University may also use, share and receive your health information in connection with this study:
  - The research sponsor and companies owned or connected with the sponsor: *The National Cancer Institute, Cancer Trials Support Unit (CTSU), Cancer Therapy Evaluation Program (CTEP), and any company supporting the study or the study agent/treatment now or in the future.*

The information that is shared with those listed above may no longer be protected by federal privacy rules.

#### **Authorization Period**

This authorization will not expire unless you change your mind and revoke it in writing. There is no set date at which your information will be destroyed or no longer used. This is because the information used and created during the study may be analyzed for many years, and it is not possible to know when this will be completed.

| Initials/Date |
|---------------|
|---------------|

#### **Signing the Authorization**

- You have the right to refuse to sign this authorization. Your health care outside of the study, payment for your health care, and your health care benefits will not be affected if you choose not to sign this form.
- You will not be able to take part in this study and will not receive any study treatments if you do not sign this form.
- If you sign this authorization, you may change your mind at any time. Researchers may continue to use information collected up until the time that you formally changed your mind. If you change your mind, your authorization must be revoked in writing. To revoke your authorization, please write to: Dr. Alice Mims, A343 Starling Loving Hall, 320 W. 10<sup>th</sup> Ave., Columbus, OH 43210. Telephone (843)-480-2685.

Or:

The HIPAA Privacy Manager, the Ohio State University Medical Center, 140 Doan Hall, 410 W. Tenth Avenue, Columbus, Ohio 43210, Telephone: (614) 293-4477.

• Signing this authorization also means that you will not be able to see or copy your study-related information until the study is completed. This includes any portion of your medical records that describes study treatment.

#### **Contacts for Questions**

- If you have any questions relating to your privacy rights, please contact: *The HIPAA Privacy Manager, the Ohio State University Medical Center, 140 Doan Hall, 410 W. Tenth Avenue, Columbus, Ohio 43210, Telephone: (614) 293-4477.*
- If you have any questions relating to the research, please contact: *Dr. Alice Mims, A343 Starling Loving Hall, 320 W. 10<sup>th</sup> Ave., Columbus, OH 43210. Telephone (843)-480-2685.*

#### **Signature**

I have read (or someone has read to me) this form and have been able to ask questions. All of my questions about this form have been answered to my satisfaction. By signing below, I permit *Dr. Alice Mims* and the others listed on this form to use and share my personal health information for this study. I will be given a copy of this signed form.

| Signature | | | |
|---|---|---|---|
| (Subject or Legally Authorized Rep | resentative) | | |
| Print Name | Date | Time | AM/PM |
| (If legal representative, also print r | elationship to subject) | | |

### **Research Study Informed Consent Document**

**Study Title for Participants:** Testing Nivolumab in combination with Decitabine and Venetoclax in Patients with Newly Diagnosed TP53 Gene Mutated Acute Myeloid Leukemia

Official Study Title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>: Protocol 10317: "A Pilot Study of Nivolumab in Combination with Decitabine and Venetoclax in *TP53*-mutated Acute Myeloid Leukemia (NCT TBD)"

### **Overview and Key Information**

### What am I being asked to do?

We are asking you to take part in a research study. This study has public funding from the National Cancer Institute (NCI), part of the National Institutes of Health (NIH) in the United States Department of Health and Human Services. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

We are asking you to take part in this research study because you have Acute Myeloid Leukemia (AML) and your cancer has a gene mutation called TP53.

### Taking part in this study is your choice.

You can choose to take part or you can choose not to take part in this study. You also can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document has important information to help you make your choice. Take time to read it. Talk to your doctor, family, or friends about the risks and benefits of taking part in the study. It's important that you have as much information as you need and that all your questions are answered. See the "Where can I get more information?" section for resources for more clinical trials and general cancer information.

### Why is this study being done?

We are doing this study because we want to find out if this approach is better or worse than the usual approach for your cancer, which is AML with TP53 gene mutation. The usual approach is defined as care most people get for AML.

One of the study drugs, called Nivolumab, is being looked at to see if it may help treat patients with your type of AML. Nivolumab works by helping your body's natural defense cells, called "T-Cells," to possibly be able to better attach to cancer cells, which then may be able to help to kill the cancer cells. Nivolumab is not currently approved by the Food and Drug Administration (FDA) for use in patients with your type of AML.

### What is the usual approach to my Acute Myeloid Leukemia (AML)?

The usual approach for patients who are not in a study is treatment with newly diagnosed AML is chemotherapy. AML patients will receive FDA approved treatment with either:

- intensive chemotherapy with two chemotherapy drugs (an anthracycline and cytarabine given together for 7 days) or
- less intensive chemotherapy (azacitidine or decitabine) without or with venetoclax (for patients age 75 and older or for patients younger who are not able to receive the intensive chemotherapy treatment).

For patients with TP53 gene mutated AML these treatments may not work well and for patients in which it does work they may have a high chance of relapse. For patients who get the usual approach for this cancer, about less than 10 out of 100 are free of cancer after 5 years.

### What are my choices if I decide not to take part in this study?

- You may choose to have the usual approach described above.
- You may choose to take part in a different research study, if one is available.
- You may choose not to be treated for cancer.
- You may choose to only get comfort care to help relieve your symptoms and not get treated for your cancer.

### What will happen if I decide to take part in this study?

If you decide to take part in this study, you will take three cancer drugs during your treatment named Decitabine, Nivolumab, and Venetoclax.

Cancer drug treatment occurs in cycles. A cycle means that you have a single cancer drug or a combination of drugs and then have a rest to allow your body to recover. Then the cycle repeats. In this study, there is a 28 day cycle, which means you will start treatment on the first day of the cycle, take the three cancer drugs as described below, then have a break at the end of the cycle before restarting all of the cancer drugs again with another cycle. At the end of each 28 day cycle, your study doctor will determine if you need to have any additional cycles of treatment.

During each cycle you will receive Decitabine on Days 1-10 for the first 3 cycles as needed, and then on days 1-5 for each subsequent cycle.

You will receive Nivolumab on Day 15 for the first cycle and on Days 1 and 15 for all of the following cycles.

You will receive Venetoclax on Days 1-21 of each cycle.

If your leukemia has not responded to treatment after three cycles, you will stop treatment. If you have responded to treatment, the treatment will be given until your health changes and the study is no longer in your best interest, you wish to stop the study, or if the study is stopped. After you finish the treatment of Decitabine, Nivolumab, and Venetoclax, your doctor will continue to follow your AML and watch you for side effects for about 3 years after you initially started this treatment combination. If you experienced any side effects, you will be followed until the side effect stop or are stable.

You will be seen by a doctor for follow up on days 1 and 15 of every cycle while you are on this study. This will continue as long as you are in the study. If you come off study, follow up will be decided by your cancer doctor.



### What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important for you to think carefully about these as you make your decision.

#### Risks

We want to make sure you know about a few key risks right now. We give you more information in the "What risks can I expect from taking part in this study?" section.

If you choose to take part in this study, there is a risk that the study drugs Decitabine, Nivolumab, and Venetoclax may not be as good as the usual approach for your cancer at putting your AML in remission.

There is also a risk that you could have side effects from the study drugs, Decitabine, Nivolumab, and Venetoclax. These side effects may be worse and may be different than you would get with the usual approach for your cancer.

Some of the most common side effects that the study doctors know about are:

- Decitabine:
  - o low white blood cell count (cells that help fight infection)
  - o low platelets (cells that help your blood clot)
- Venetoclax:
  - o low white blood cell count (cells that help fight infection)
  - o Tumor Lysis Syndrome (TLS) which a serious and life threatening condition
- Nivolumab:
  - A severe immune response which may attack your organs such as your skin, lungs, intestines, kidneys, liver and other organs within your body. These immune responses can be severe and possibly fatal

There may be some risks that the study doctors do not yet know about.

#### **Benefits**

There is some evidence with AML that adding Nivolumab to Decitabine and Venetoclax to the usual approach may stabilize cancer for longer than the usual approach alone, and may put the cancer in remission more frequently than the usual approach alone. However, we do not know if this will happen in people with TP53 gene mutated AML. It is unlikely that this Nivolumab with Dectabine and Venetoclax will help you live longer than the usual approach alone. This study may help the study doctors learn things that may help other people in the future.

### If I decide to take part in this study, can I stop later?

Yes, you can decide to stop taking part in the study at any time.

If you decide to stop, let your study doctor know as soon as possible. It's important that you stop safely. If you stop, you can decide if you want to keep letting the study doctor know how you are doing.

Your study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

### Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:

- Your health changes and the study is no longer in your best interest.
- New information becomes available and the study is no longer in your best interest.

- You do not follow the study rules.
- For women: You become pregnant while on the study.
- You complete a bone marrow/stem cell transplantation
- The study is stopped by the Institutional Review Board (IRB), Food and Drug Administration (FDA), or study sponsor, The National Cancer Institute (NCI) the study sponsor. The study sponsor is the organization who oversees the study.

It is important that you understand the information in the informed consent before making your decision. Please read, or have someone read to you, the rest of this document. If there is anything you don't understand, be sure to ask your study doctor or nurse.

### What is the purpose of this study?

The purpose of this study is to test the safety of a combination of chemotherapy drugs called Nivolumab, Decitabine, and Venetoclax. These drugs are not approved by the FDA to treat patients with TP53 gene mutated AML. There will be about 15 people taking part in this study.

The mutation in this study being testing is the TP53 (tumor protein) gene mutation. This protein helps stop the growth of tumors. In order to participate in this study you must have AML with the TP53 gene mutation. To determine if you have this mutation an extra tube of blood will be drawn at the time of screening and a bone marrow aspirate will be completed.

### What are the study groups?

This study has a screening step. The purpose of this step is to test your tumor to find out if it has a specific mutation. If it does and you meet all the study requirements, then we can assign you to treatment based on these changes. If we find that your blood or bone marrow aspirate does not have the mutation that is needed for this study, then your doctor will discuss other options for your care. This screening test is not approved by the FDA for your AML.

All patients in this study will receive the chemotherapy combination Decitabine, Nivolumab, and Venetoclax in 28 day cycles until your health changes and the study is no longer in your best interest, you wish to stop the study, or if the study is stopped.

During each cycle you will receive Decitabine (20mg/m²) through a vein in your arm for approximately 60 minutes on Days 1-10 for up to the first 3 cycles as needed and then on days 1-5 for each subsequent cycle.

You will receive Nivolumab (240 mg) through a vein in your arm for approximately 30 minutes on Day 15 for the first cycle and on Days 1 and 15 for all subsequent cycles.

You will take Venetoclax by mouth with food and water on Days 1-21 of each cycle. During cycle 1 you will take 100mg on Day 1, 200mg on Day 2, and 400 mg on Days 3-21. After cycle

1 you will take 400mgs on Days 1-21. If you are taking certain medications that can interact with Venetoclax, this dosing may be adjusted.

You will be able to get additional doses of the Decitabine and Venetoclax if appropriate, as these are approved by the FDA for treatment of your disease. You will not be able to get additional doses of the Nivolumab. This drug is not approved by the FDA for treatment of your disease.

### What exams, tests, and procedures are involved in this study?

Before you begin the study, your doctor will review the results of your exams, tests, and procedures. This helps your doctor decide if it is safe for you to take part in the study. If you join the study, you will have more exams, tests, and procedures to closely monitor your safety and health. Most of these are included in the usual care you would get even if you were not in a study.

Listed below are exams, tests, and procedures that need to be done as part of this study to monitor your safety and health, but may not be included in the usual care. We will use them to carefully follow the effects of the study treatment, including preventing and managing side effects.

These exams, tests, and procedures to monitor your safety and health include:

- Blood counts (will check your levels to determine risk of infection and if needs for blood or platelet transfusions):
  - o screening
  - twice weekly during first cycle of induction and during cycles 2-3 of induction if these cycles are needed
  - o Day 1 of each cycle of maintenance
  - o when stopping study treatment
- Blood testing (to check your electrolytes and your organ function of kidneys and liver
  - screening
  - o every 12 hours during the first 4 days of venetoclax during cycle 1
  - o twice weekly during first cycle of induction and during cycles 2-3 of induction if these cycles are needed
  - O Day 1 of each cycle of maintenance
  - o when stopping study treatment
- A set of questions to determine how well you can complete your daily activities
  - o screening
  - o Day 1 of every cycle
  - when stopping study treatment
- Physical exams
  - o screening
  - O Days 1 and 15 of every cycle
  - o when stopping study treatment
- Bone Marrow biopsy for AML cells and genetic testing at

- o screening
- End of first cycle of induction and end of cycles 2-3 of induction if these cycles are needed
- o every 3 cycles during maintenance cycles a
- o when stopping study treatment

This study will use genetic tests that may identify changes in the genes in your tumor DNA. Your genes carry information about you and your family, from the color of your eyes to health conditions for which you may be at risk, such as certain kinds of cancer.

Finding these changes would not affect your treatment in this study. However, they could affect your health in other ways. If there are changes found that could cause health problems, then your study doctor will discuss your options with you. As appropriate, you may be referred for genetic counseling.

Some exams, tests, and procedures are a necessary part of the research study, but would not be included in usual care. Listed below are procedures that will be done for research purposes only.

You will need to have blood and bone marrow samples taken for the study at screening and at the end of each cycle of treatment. These samples will be used for research purposes to look at other features of your leukemia cells that may help determine how to better target leukemia cells with treatment for future patients with TP53 gene mutations. You and your study doctor will not get the results of this testing. If you agree to take part in the study, you may need to sign a separate consent form for the study biopsy at the hospital or clinic where the biopsy is done.

Your study doctor will need to draw some extra liquid during your bone marrow biopsies at screening and after cycles 1-3 and every 3 cycles until the end of treatment. The sample at screening will determine if you have a TP53 gene mutation and other samples will be used for exploratory biomarkers for research purposes to look at other features of your leukemia cells that may help determine how to better target leukemia cells with treatment for future patients with TP53 gene mutations. You and your study doctor will get the results of the TP53 gene mutation testing but will not get results of other research testing.

Please see the optional research sample section for information regarding the optional research studies.

### What risks can I expect from taking part in this study?

#### **General Risks**

If you choose to take part in this study, there is a risk that the addition of Nivolumab given with Venetoclax and Decitabine may not be as good as the usual approach for your AML at getting it into remission.

You also may have the following discomforts:

- Spend more time in the hospital or doctor's office.
- Be asked sensitive or private questions about things you normally do not discuss.
- May not be able to take part in future studies.

The Nivolumab, Decitabine, and Venetoclax used in this study could be very harmful to an unborn or newborn baby. There may be some risks that doctors do not yet know about. It is very important that you check with your study doctor about what types of birth control or pregnancy prevention to use during the study and for 7 months for men and 6 months for women after you have completed the study.

#### **Genetic Testing Risks**

The genetic test used in this study will test your tumor for a gene mutation called TP53. This change also may be in your normal tissue and passed down through your family. For example, these genetic changes may be passed down to your children in the same way that eye and hair color are passed down.

Since this study is only testing tumor tissue, we will not know if a genetic change in your tumor is also in your normal tissue. If you want to find out if the change is in your normal tissue, then you will need to get other tests done outside of this study.

Genetic tests of normal tissue can reveal information about you and also about your relatives. Your study doctor will talk with you about what testing your normal tissue may mean for you and your family. He or she also may suggest that you talk with a genetics counselor to learn more. You or your insurance plan would have to pay for any genetic tests and visits to a genetic counselor done outside of this study.

#### **Biopsy Risks**

Common side effects of a biopsy are a small amount of bleeding at the time of the procedure, bruising, and pain at the biopsy site. Pain can be treated with regular pain medications. Rarely, an infection can occur. You may sign a separate consent form for the study biopsy that describes the risks in more detail.

#### **Side Effect Risks**

The drugs used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will test your blood and let you know if changes occur that may affect your health.

Here are important things to know about side effects:

- 1. The study doctors do not know who will or will not have side effects.
- 2. Some side effects may go away soon, some may last a long time, and some may never go away.

3. Some side effects may be mild. Other side effects may be very serious and even result in death.

You can ask your study doctor questions about side effects at any time. Here are important ways to make side effects less of a problem:

- If you notice or feel anything different, tell your study doctor. He or she can check to see if it is a side effect.
- Your study doctor will work with you to treat your side effects.
- Your study doctor may adjust the study drugs to try to reduce side effects.

This study is looking at a combination of the usual drugs used to treat this type of cancer plus a study drug. This different combination of drugs may increase your side effects or may cause new side effects.

There is also a risk that you could have other side effects from the study such as side effects from the blood draws and bone marrow biopsies.

#### **Drug Risks**

The tables below show the most common and most serious side effects doctors know about. Keep in mind that there might be other side effects doctors do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

#### **Possible Side Effects for Decitabine**

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving decitabine (5-aza-2'-deoxycytidine), more than 20 and up to 100 may have:

- Anemia, which may require blood transfusion
- Nausea
- Tiredness, fever
- Infection, especially when white blood count is low
- Bruising, bleeding

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving decitabine (5-aza-2'-deoxycytidine), from 4 to 20 may have:

- Pain
- Constipation, diarrhea, vomiting
- Sores in the mouth which may cause difficulty swallowing
- Chills
- Swelling of the body
- Damage to the body by own immune system
- Loss of appetite
- Dizziness, headache
- Worry

- Difficulty sleeping
- Cough, shortness of breath, sore throat
- Internal bleeding which may cause coughing up blood
- Bleeding from multiple sites including the nose
- Hair loss, itching, rash

#### RARE, AND SERIOUS

In 100 people receiving decitabine (5-aza-2'-deoxycytidine), 3 or fewer may have:

• Bleeding in the brain which may cause confusion

Possible Side Effects of Nivolumab (Table Version Date: June 18, 2018)

#### PLEASE NOTE THE FOLLOWING IN REVIEWING THESE RISKS:

BMS-936558 (nivolumab) is an agent involved in the inhibition of "immune checkpoints," and may result in severe and possibly fatal immune-mediated side effects probably due to activation and growth of immune cells (T-cells). Immune-mediated side effects have been reported in patients receiving BMS-936558 (nivolumab). In clinical trials, most immune-mediated side effects were reversible and managed by stopping BMS-936558 (nivolumab) temporarily, administration of corticosteroids, and supportive care.

#### **Special precautions**

Side effects of BMS-936558 (nivolumab, MDX-1106) may happen anytime during treatment or even after your treatment has ended. Some of these problems may happen more often when BMS-936558 (nivolumab, MDX-1106) is used in combination with ipilimumab. Call or see your healthcare provider right away if you develop any problems listed below or the symptoms get worse.

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving BMS-936558 (nivolumab, MDX-1106), more than 20 and up to 100 may have:

Tiredness

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving BMS-936558 (nivolumab, MDX-1106), from 4 to 20 may have:

- Anemia, which may require blood transfusion
- Swelling and redness of the eye
- Pain
- Diarrhea or nausea
- Dry mouth
- Fever
- Swelling and redness at the site of the medication injection
- Bruising or bleeding

- Pain or swelling of the joints
- Loss of appetite
- Reaction during or following a drug infusion which may cause fever, chills, or rash

BMS-936558 (nivolumab, MDX-1106) may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:

- Lung problems (pneumonitis and pleural effusion). Symptoms may include: new or worsening cough, chest pain, or shortness of breath.
- Intestinal problems (colitis) that can rarely lead to tears or holes in your intestines. Signs and symptoms of colitis may include: diarrhea or increase in bowel movements; blood in your stools or dark, tarry, sticky stools; severe belly pain or tenderness.
- Skin problems, including itching; rash, blisters including on the inside the mouth; or loss of skin pigment
- Liver problems (hepatitis) which can cause liver failure. Signs and symptoms of hepatitis may include: yellowing of your skin or the whites of your eyes, severe nausea or vomiting, drowsiness, or pain in the right upper belly
- Hormone gland problems (especially the thyroid, pituitary and adrenal glands, and pancreas). Signs and symptoms may include: headaches that will not go away or unusual headaches; extreme tiredness, or changes in mood or behavior; decreased sex drive; weight loss or weight gain; excessive thirst or urine; or dizziness or fainting.

### RARE, AND SERIOUS

In 100 people receiving BMS-936558 (nivolumab, MDX-1106), 3 or fewer may have:

- Dry eyes
- Sores in the mouth which may cause difficulty swallowing

BMS-936558 (nivolumab, MDX-1106) may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:

- Visual disturbances which may cause double vision, blurred vision, or loss of vision with a chance of blindness
- A condition with high blood sugar which leads to tiredness, frequent urination, excessive thirst, headache, nausea and vomiting, and can result in coma
- Kidney problems, including nephritis and kidney failure requiring dialysis. Signs
  of kidney problems may include decrease in the amount of urine, blood in your
  urine, or ankle swelling.
- Heart problems, including swelling and heart failure. Symptoms and signs of heart problem may include shortness of breath, or swelling of the ankle and body.
- Muscle problems, including swelling, which can cause muscle pain and severe muscle weakness, sometimes with dark urine

- Swelling of the brain (meningitis/encephalitis) which may cause headaches; stiff neck; confusion; sleepiness; seizures; injury to the brain; or blindness (also known as Reversible Posterior Leukoencephalopathy Syndrome)
- Nerve problems that can cause paralysis. Signs and symptoms may include numbness; tingling of hands and feet; weakness of the arms, legs, and facial muscle movements
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, or swelling of the face or throat
- Complications associated with stem cell transplant using donor stem cells (allogeneic stem cell transplant). These complications are caused by attack of donor cells on the host organs (inducing liver, skin, and gut damage), and can lead to death. If you are considering an allogeneic stem transplant after participating in this study, please tell your doctor that you have received nivolumab therapy, since the risk and severity of transplant-associated complications may be increased.

#### Possible Side Effects of Venetoclax (ABT-199):

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving venetoclax (ABT-199), more than 20 and up to 100 may have:

- Anemia, which may require blood transfusion
- Diarrhea, nausea
- Tiredness
- Infection, especially when white blood cell count is low

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving venetoclax (ABT-199), from 4 to 20 may have:

- Constipation, vomiting
- Fever
- Bruising, bleeding
- Pain in joints
- Headache
- Cough
- High blood pressure which may cause headaches, dizziness, blurred vision

#### RARE, AND SERIOUS

In 100 people receiving venetoclax (ABT-199), 3 or fewer may have:

Kidney damage which may require dialysis

#### **Additional Drug Risks**

The study drugs could interact with other drugs. If you are taking other drugs that suppress your immune system, the addition of Nivolumab may make this worse.

Rarely, there are problems getting enough supplies of the Nivolumab. If that happens, your doctor will talk with you about your options.

### What are my responsibilities in this study?

If you choose to take part in this study you will need to:

- Keep your study appointments.
- Write down in your medication diary when you take the study drug at home Tell your doctor about:
  - o all medications and supplements you are taking
  - o any side effects
  - o any doctors' visits or hospital stays outside of this study
  - o if you have been or are currently in another research study.

**For women:** Do not get pregnant or breastfeed while taking part in this study. **For men:** Do not father a baby while taking part in this study. **For all:** Tell your study doctor right away if you think that you or your partner have become pregnant during the study or within 7 months for men and 6 months for women after your last day of study treatment.

### What are the costs of taking part in this study?

You and/or your insurance plan will need to pay for the costs of medical care you get as part of the study, just as you would if you were getting the usual care for your cancer. This includes:

- the costs of tests, exams, procedures, and drugs that you get during the study to monitor your safety, and prevent and treat side effects.
- the costs of getting the IV drugs ready and giving them to you.
- your insurance co-pays and deductibles.

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it doesn't pay for if you take part in this clinical trial. Also, find out if you need approval from your plan before you can take part in the study.

Ask your doctor or nurse for help finding the right person to talk to if you are unsure which costs will be billed to you or your insurance provider.

You and/or your insurance provider will not have to pay for exams, tests, and procedures done for research purposes only or that are covered by the study. These include:

- The extra blood samples and bone marrow biopsy samples taken for research.
- The time points at which each blood sample and bone marrow biopsy will occur are:
  - O During screening: blood and bone marrow
  - O Day 28 +/- 1 day of cycles 1, 2, and 3: blood and bone marrow
  - O Day 28 +/- 1 day every 3 cycles starting with cycle 6 (ex. Cycles 6, 9, 12...): blood and bone marrow
  - Day 28 +/- 1 day of end of every cycle starting with cycle 4 (excluding cycles 6,9, 12...as above): blood only
  - o End of Treatment or AML Relapse: blood and bone marrow

You or your insurance provider will not have to pay for the Nivolumab drug itself while you take part in this study.

Taking part in this study may mean that you need to make more visits to the clinic or hospital than if you were getting the usual approach to treat your cancer. You may:

- Have more travel costs.
- Need to take more time off work.
- Have other additional personal costs.

You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

### What happens if I am injured because I took part in this study?

If you are injured as a result of taking part in this study and need medical treatment, please talk with your study doctor right away about your treatment options. The study sponsors will not pay for medical treatment for injury. Your insurance company may not be willing to pay for a study-related injury. Ask them if they will pay. If you do not have insurance, then you would need to pay for these medical costs.

If you feel this injury was caused by medical error on the part of the study doctors or others involved in the study, you have the legal right to seek payment, even though you are in a study. Agreeing to take part in this study does not mean you give up these rights.

The Ohio State University has no funds set aside for the payment of health care expenses for this study.

### Who will see my medical information?

Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are.

Some of your health information, such as your response to cancer treatment, results of study tests, and medicines you took, will be kept by the study sponsor in a central research database. However, your name and contact information will not be put in the database. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

There are organizations that may look at or receive copies of some of the information in your study records. Your health information in the research database also may be shared with these organizations. They must keep your information private, unless required by law to give it to another group.

#### Some of these organizations are:

- The study sponsor and any company supporting the study or the study agent/treatment now or in the future. This would include any organization helping the company with the study.
- The National Cancer Institute (NCI) Central Institutional Review Board (CIRB), which is a group of people who review the research with the goal of protecting the people who take part in the study.
- The Food and Drug Administration (FDA) and the groups it works with to review research.
- The National Cancer Institute (NCI) and the groups it works with to review research.
- The NCI's National Clinical Trials Network and the groups it works with to conduct research
- The Ohio State University researchers and staff, who may share or use health information about you with others involved in this study. For example, this may include your medical and research records, any imaging tests or scans such as x-rays, and laboratory results.

In addition to storing data in the study database, data from studies that are publicly funded may also be shared broadly for future research with protections for your privacy. The goal of this data sharing is to make more research possible that may improve people's health. Your study records may be stored and shared for future use in public databases. However, your name and other personal information will not be used.

Some types of future research may include looking at your information and information from other patients to see who had side effects across many studies or comparing new study data with older study data. However, right now we don't know what research may be done in the future using your information. This means that:

- You will not be asked if you agree to take part in the specific future research studies using your health information.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your information.

There are laws that protect your genetic information. However, there is a risk that someone could get access to your genetic information and identify you by name. In some cases, employers could use your genetic information to decide whether to hire or fire you. The study doctors believe the risk of this happening is very small. However, the risk may increase in the future as people find new ways of tracing information. For more information about the laws that protect you, ask your study doctor.

### Where can I get more information?

You may visit the NCI web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can talk to the study doctor about any questions or concerns you have about this study or to report side effects or injuries. Contact the study doctor, Alice Mims, MD at 614-685-6031 or Alice.Mims@osumc.edu.

For questions about your rights while in this study, call Ms. Sandra Meadows in The Office of Responsible Research Practices at 1-800-678-6251.

### Optional studies that you can choose to take part in

This part of the consent form is about optional studies that you can choose to take part in. They are separate from the main study described above. These optional studies will not benefit your health. The researchers leading these optional studies hope the results will help other people with cancer in the future. The results will not be added to your medical records and you or your study doctor will not know the results.

Taking part in these optional studies is your choice. You can still take part in the main study even if you say "no" to any or all of these studies. There is no penalty for saying "no." You and your insurance company will not be billed for these optional studies. If you sign up for, but cannot complete any of these studies for any reason, you can still take part in the main study.

Circle your choice of "yes" or "no" for each of the following studies.

## Optional sample collections for known laboratory studies and/or storage for possible future studies

Researchers are trying to learn more about cancer and other health problems using blood and tissue samples from people who take part in clinical trials. By studying these samples, researchers hope to find new ways to prevent, detect, treat, or cure diseases.

Some of these studies may be about how genes affect health and disease. Other studies may look at how genes affect a person's response to treatment. Genes carry information about traits that are found in you and your family. Examples of traits are the color of your eyes, having curly or straight hair, and certain health conditions that are passed down in families. Some of the studies may lead to new products, such as drugs or tests for diseases.

#### **Known future studies**

If you choose to take part in this optional study, researchers will collect blood and bone marrow for research on leukemia cells with TP53 gene mutations. Your samples will be used for to look at other features of your leukemia cells (besides the TP53 gene mutation) that may help determine how to better target leukemia cells with treatment for future patients with TP53 gene mutations.

Your study doctor will need to draw some extra liquid during your bone marrow biopsies at screening and after cycles 1-3 and every 3 cycles until the end of treatment. The sample at screening will determine if you have a TP53 gene mutation and other You and your study doctor will get the results of the TP53 gene mutation testing but will not get results of other research testing.

#### What is involved in this optional sample collection?

If you agree to take part, here is what will happen next:

1. About <sup>3</sup>/<sub>4</sub> tablespoons of blood will be collected from a vein in your arm (this is from the blood draw you are already getting as part of the study). A sample of bone marrow will be collected from a biopsy (this is from the biopsies you are already getting as part of the study, and is not a separate collection of your bone marrow).

#### What are the risks in this optional sample collection?

- The most common risks related to drawing blood from your arm are brief pain and maybe a bruise.
- The most commons risks related to bone marrow biopsies are brief pain and maybe a bruise.
- Your medical and genetic information is unique to you. There is a risk that someone
  outside of the research study could get access to your study records or trace information
  in a database back to you. They could use that information in a way that could harm you.
  Researchers believe the chance that someone could access and misuse your information is
  very small. However, the risk may increase in the future as people find new ways of
  tracing information.

#### How will information about me be kept private?

Your privacy is very important to the study researchers and biobank. They will make every effort to protect it. Here are just a few of the steps they will take:

- 1. They will remove identifiers, such as your initials, from your sample and information. They will replace them with a code number. There will be a master list linking the code numbers to names, but they will keep it separate from the samples and information.
- 2. Researchers who study your sample and information will not know who you are. They also must agree that they will not try to find out who you are.
- 3. Your personal information will not be given to anyone unless it is required by law.
- 4. If research results are published, your name and other personal information will not be used.

#### What are the benefits to taking part in this optional sample collection?

You will not benefit from taking part.

The researchers, using the samples from you and others, might make discoveries that could help people in the future.

#### Are there any costs or payments to this optional sample collection?

There are no costs to you or your insurance. You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

#### What if I change my mind about this optional sample collection?

If you decide you no longer want your samples to be used, you can call the study doctor, Alice Mims, MD at 843-480-2685, who will let the rest of the study team know. Then, any sample that remains will be destroyed or returned to your study doctor. This will not apply to any samples or related health information that have already been given to or used by researchers.

#### What if I have questions about this optional sample collection?

If you have questions about the use of your samples for research, contact the study doctor, Alice Mims, MD at 843-480-2685.

Please circle your answer below to show if you would or would not like to take part in each optional study:

### Samples for known future studies:

I agree that my samples and related health information may be used for the laboratory (\*study or studies\*) described above.

YES NO

This is the end of the section about optional studies.

### My signature agreeing to take part in the study

I have read this consent form or had it read to me. I have discussed it with the study doctor and my questions have been answered. I will be given a signed and dated copy of this form. I agree to take part in the main study.

| Participant's sign | ature | | |
|---|---|---|---|
| Date of signature _ | | | |
| Time | AM/PM | | |
| Signature of perso | on(s) conducting the info | ormed consent discussion | |
| Date of signature | | | |
| Time | AM/PM | | |
| <u>Witness(es)</u> [As ар | oplicable to the research] | | |
| Printed nam | ne of witness | Signature of witness | |
| | | | AM/PM |
| | | Date and time | |